CLINICAL TRIAL: NCT05645315
Title: A Phase Ib Clinical Trial to Evaluate the Efficacy and Safety of TQB2618 Injection Combined With TQB2450 Injection in Patients With Advanced Solid Tumors
Brief Title: Clinical Trial of TQB2618 Injection Combined With TQB2450 Injection in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2618-TQB2450-Ib-01
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2618 injection+TQB2450 injection (Experimental): TQB2618 injection combined with TQB2450 injection, 21 days as a treatment cycle.
  Interventions: Drug: TQB2618 injection and TQB2450 injection

INTERVENTIONS:
Drug: TQB2618 injection and TQB2450 injection — TQB2618 is a TIM-3 receptor monoclonal antibody; TQB2450 is a new sequence of innovative anti-PD-L1 fully humanized monoclonal antibody;

SUMMARY:
This project is a phase Ib clinical trial study evaluating the efficacy and safety of TQB2618 injection combined with TQB2450 injection in patients with advanced solid tumors, the trial plan to enroll 127 subjects, the trial design is a phase I.b dose exploration and cohort expansion clinical study, aiming to evaluate the safety and efficacy of TQB2618 injection combined with TQB2450 injection in patients with advanced malignant solid tumors, and to evaluate TQB2618 injection, Pharmacokinetic characteristics, receptor occupancy and immunogenicity characteristics of TQB2450 injection; Biomarker studies related to the mechanism of action, safety and/or pathological mechanism of efficacy have dose-limiting toxicity (DLT) in Phase I, recommended dose in Phase II (RP2D), and objective response rate (ORR) in Phase II as the primary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* The subjects voluntarily participated the study and signed the informed consent form;
* Age: 18~75 years old (when signing the informed consent form); ECOG PS score: 0~1 points; Expected survival is more than 3 months;
* The enrolled patients meet the following criteria:

  1. Satge I (dose exploration): patients with advanced malignant solid tumors confirmed by tissue and/or cytology, where standard therapy has failed or there is a lack of effective treatment;
  2. Stage 2 (cohort Expansion):

     1. Cohort 1: PD-L1-positive patients with advanced first-line NSCLC;
     2. Cohort 2: PD-L1 positive patients with advanced immunoresistant NSCLC;

        1. Patients with locally advanced (stage III.B/III.C), recurrent or metastatic (stage IV) NSCLC who are not histologically or cytologically confirmed and are not suitable for radical concurrent chemoradiotherapy.
        2. For non-squamous non-small cell lung cancer, the test proves the absence of EGFR mutation, ALK fusion, ROS1 mutation (for squamous non-small cell lung cancer, patients with known mutations in the above genes are excluded, and testing is not mandatory for those whose status is unknown);
        3. Positive PD-L1 expression ratio≥1% [TC (tumor cells) or IC (immune cells) ≥1%];
        4. Cohort 1 advanced first-line patients: no systemic antitumor therapy for advanced disease.
        5. Patients with advanced immunoresistance in cohort 2: at least prior failure of platinum-containing chemotherapy and immune checkpoint inhibitor (PD-1 or PD-L1) therapy (combined or sequential therapy allowed)
* at least one measurable lesion confirmed according to RECIST 1.1;
* The main organs function normally
* Female subjects of childbearing age should agree that contraception must be used during the study and for 6 months after the end of the study

Exclusion Criteria:

* Comorbidities and medical history:

  1. Have received chemotherapy within 3 weeks before the first dose, radiotherapy (except palliative radiotherapy for non-target lesions) or other antineoplastic drugs within 2 weeks before the first dose (the washout period is calculated from the end of the last treatment);
  2. Have developed or are currently suffering from other malignant tumors within 3 years before the first dose. The following two conditions can be enrolled: other malignancies treated with a single surgery, achieving 5 consecutive years of disease-free survival (DFS); cured carcinoma in situ, non-melanoma skin cancer, and superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ), and T1 (tumor-invasive basement membrane)];
  3. unresolved toxicities above CTC AE grade 1 due to any prior treatment, excluding hair loss;
  4. Major surgical treatment and obvious traumatic injury within 28 days before the first dose;
  5. Wounds or fractures that have not healed for a long time;
  6. Arterioven/venous thrombotic events within 6 months prior to the first dose;
  7. Those with a history of psychotropic substance abuse and cannot quit or have mental disorders;
  8. Subjects with any severe and/or uncontrolled disease.
* Tumor-related symptoms and treatment:

  1. Received proprietary Chinese medicine treatment with anti-tumor indications specified in the NMPA-approved drug instructions within 2 weeks before the first dose;
  2. Have received previous anti-TIM-3 antibody treatment;
  3. Have received previous immunotherapy drugs such as anti-PD-1/PD-L1 antibody and anti-CTLA-4 antibody (only applicable to cohort 1 of the Stage II cohort expansion study: advanced first-line NSCLC patients with positive PD-L1 expression);
  4. uncontrolled pleural effusion, pericardial effusion, or ascites that still requires repeated drainage (judged by the investigator);
  5. Known spinal cord compression, cancerous meningitis, with symptoms of brain metastases or symptom control for less than 2 weeks;
* Study treatment-related:

  1. History of live attenuated vaccination within 28 days before the first dose or planned live attenuated vaccination during the study period;
  2. Those who have severe hypersensitivity reactions after using macromolecular drugs;
  3. Active autoimmune disease requiring systemic therapy within 2 years before the first dose (e.g., use of disease-modifying drugs, corticosteroids, or immunosuppressants); asthma patients requiring bronchodilators for medical intervention.
* Those who have participated in and used other anti-tumor clinical trial drugs within 4 weeks before the first dose;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity | within the first treatment cycle for 21 days
  The occurrence of severe toxicities during the first cycle of anti-cancer therapy
Phase II recommended dose | Through phase 1 completion, an average of half a year
  Dose selection in the expansion phase
Objective response rate | Up to 12 months
  ORR is defined as the percentage of participants with progressive disease (PD) from first dose to first recorded or death from any cause of complete remission (CR) and partial remission (PR) based on investigator records

SECONDARY OUTCOMES:
Progression-free survival | Up to 12 months
  PFS is defined as the time from randomization to the first recorded progressive disease (PD) or death from any cause.
Disease control rate | Up to 12 months
  The time when participants first achieved full or partial remission of disease progression.
Duration of remission | Up to 12 months
  The time from the start of the first evaluation of the tumor as Complete Response or Partial Response to the first assessment as Progressive Disease or death from any cause.
Overall survival | Up to 18 months
  OS is defined as the time from randomization to death from any cause. Participants who did not die at the end of the extended follow-up period, or who lost follow-up during the study, were reviewed on the last date known to be alive.
Maximum plasma drug concentration | 1 hour before and 30 minutes after TQB2450 injection administration; 30 minutes, 4, 8, 24, 48, 144, 312 hours after TQB2618 injection administration of cycle 1; 30 minutes after TQB2618 injection administration of cycle 2-8. Each cycle is 21 days.
  Maximum plasma drug concentration ia a pharmacokinetic parameter
Immunogenicity | Each cycle is 21 days. 1 hour before administration of cycles 1, 2, 4, and 8, 1 hour before administration at the start of every 6 cycles thereafter; 30 and 90 days after the last dose.
  Immunogenicity is evaluated by the detection of anti-drug antibodies (ADA) after administration
Free Tim3 receptors on the surface of CD3+ T cells | before and 30 minutes after the end of administration of per cycle during cycles 1-8; when patients withdrawn from the group due to Progression Disease
  TIM-3 receptor mass (RO) of TQB2618 on human immune cell membranes
Adverse events (AEs) | Up to 28 days after last dose or the initiation of a new antineoplastic therapy, whichever comes first
  Occurrence rate of all adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Tongji Hospital,Tongji Medical College of HUST, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - West China Hospital of Sichuan University, Chengdu, Sichuan